CLINICAL TRIAL: NCT05042960
Title: Investigating the Effects of Screen Brightness and Warm Tone Modulation on Dry Eye Symptoms
Brief Title: Computer Screen Properties Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-00472
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Light Pollution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 50% brightness group (Experimental): Participants will be using a computer screen reducing screen brightness 50%.
  Interventions: Other: Brightness
- Light App group (Experimental): Participants in this group will use a modulating computer screen tone with flux or night shift app.
  Interventions: Other: Brightness
- Control group (No Intervention): Participants in this group will be a control with no change in screen features

INTERVENTIONS:
Other: Brightness — Changing the colors or brightness on the device (computer screen) for one month
  Arms: 50% brightness group; Light App group

SUMMARY:
The purpose of this study is to identify how various popular methods of changing computer screen settings affect dry eye symptoms (eye pain, grittiness, tearing, burning, etc.). Specifically, this study will examine if there are differences in effects of blue light blocking (F.lux app or night shift) versus reducing screen brightness on the symptoms of dry eye.

DETAILED DESCRIPTION:
After the initial survey, participants will be randomized by a randomization tool internal to Redcap to be in one of three arms of intervention: no intervention, screen brightness reduction to 50%, and tone modulator application. Instructions will be e-mailed to participants to explain the steps they must take depending on which treatment arm they are randomized to. Adherence will be monitored and assessed at the time of post-intervention survey. If participants have issues with the software of complying, they will be able to contact the research team at any point.

ELIGIBILITY:
Inclusion Criteria:

* Adult person (18+) with intact vision who uses computers

Exclusion Criteria:

* Children (<18 years)
* Adult person without intact vision
* Adult who does not use computer screens

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
The frequency of dry eye symptoms | Day 1
  Participants will complete a pre-intervention survey to measure the frequency of dry eye symptoms.
The frequency of dry eye symptoms | Day 30
  Participants will complete a post-intervention survey to measure the frequency of dry eye symptoms.
The severity of dry eye symptoms | Day 1
  Participants will complete a pre-intervention survey to measure the severity of dry eye symptoms.
The severity of dry eye symptoms | Day 30
  Participants will complete a post-intervention survey to measure the severity of dry eye symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Leela Raju, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Requests should be directed to sachi.patil@nyulangone.org To gain access, data requestors will need to sign a data access agreement. Researchers who provide a methodologically sound proposal.Upon reasonable request